CLINICAL TRIAL: NCT00164424
Title: Impact of Episodic Acyclovir Therapy on Ulcer Duration and HIV Shedding From Genital Ulcers Among Men in South Africa
Brief Title: Episodic Acyclovir Therapy for Genital Ulcers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: London School of Hygiene and Tropical Medicine (Other); National Institute for Communicable Diseases, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-4294
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Ulcer; Herpes Simplex
Keywords: HSV2; genital ulcer; HIV; South Africa; Treatment; Acyclovir; Prevention
MeSH Terms: conditions — HIV Infections; Ulcer; Herpes Simplex | interventions — Acyclovir

INTERVENTIONS:
Drug: Acyclovir

SUMMARY:
The purpose of this study is to determine if acyclovir episodic treatment has an effect in ulcer healing and if it should be added to the syndromic management of genital ulcer disease.

DETAILED DESCRIPTION:
Background and Objectives: Herpes simplex virus type 2 (HSV-2) is the primary cause of genital ulcer and one of the most prevalent sexually transmitted infections (STI) worldwide. HSV-2 has been recognized as a risk factor for HIV in multiple studies. A substantial shift in the aetiology of genital ulcer disease (GUD) towards genital herpes has been noted in many countries in Africa, especially those with mature HIV epidemics. Some countries guided by the predominance of HSV-2 as the aetiology of GUD in their country, are changing syndromic guidelines to include acyclovir as part of the treatment for GUD. Little data is available to support this decision in terms of its effect on clinical course and its cost-effectiveness. Yet, substantial investment would be needed in poor countries to add acyclovir to their essential drug list. Studies to determine the appropriateness of episodic acyclovir therapy for HSV-2 in the developing world are needed.

Episodic therapy with acyclovir both as a treatment modality and as an HIV-prevention strategy is appealing, in terms of cost and sustainability. However, it is not clear which will be its impact under field conditions in which there would be delay in symptom recognition and treatment initiation, and whether these conditions could be optimized through patient education. We propose to conduct a randomized placebo-controlled trial of the effect of HSV-2 episodic therapy on symptomatic herpes and on HIV shedding from genital ulcers. This study will help answer the question if acyclovir therapy for herpes should be added into the syndromic management of genital ulcer disease. Acyclovir has an acceptable profile for widespread STI treatment and is now relatively inexpensive and well-tolerated. Given that HSV-2 is the leading cause of GUD in the developing world, this approach could have great public health importance, by providing a safe, acceptable, and cost-effective method to treat genital ulcer disease and potentially reduce HIV transmission. If acyclovir therapy reduces HIV shedding, its incorporation into syndromic management would provide and effective way to scale it up as a public health intervention.

Methods: We plan an individually randomized double blind placebo-control trial of the WHO and US CDC recommended dose of 3-times daily acyclovir for a 5-day treatment course. The trial will be conducted at two primary health care clinics in Johannesburg, South Africa. A total of 600 men presenting to the clinic with GUD will be enrolled in the study. Consenting participants will be randomized to receive either acyclovir plus syndromic management or placebo plus syndromic management. Syndromic management for genital ulcer disease will consist of one dose antibiotics to cover for syphilis and chancroid. Participants will be followed for a month; during follow-up visits duration of ulcers, ulcer number and size will be evaluated and ulcer, blood and semen samples collected to test for HIV RNA viral loads among HIV-positives and for HSV-2 shedding.

Timeline: Duration of the project is 2 years

Expected Outcomes: The main outcome of the study will be the evaluation of the impact of acyclovir therapy on ulcer healing. We will also measure the impact of acyclovir therapy on HIV and HSV-2 viral load from genital ulcers and HIV viral load in semen.

ELIGIBILITY:
Inclusion Criteria:

* Males presenting at the primary health care clinic with a genital ulcer
* Age 18 years or older
* Willing and able to give informed consent
* Willing to be tested for HSV and HIV
* Willing and able to comply with the study protocol including follow-up visits
* Willing to accept therapy by chance

Exclusion Criteria:

* Extensive ulceration
* Ulceration >1 month
* History of adverse reaction to acyclovir
* Taking suppressive therapy for genital herpes
* History of renal insufficiency or proteinuria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2005-03; Primary Completion 2009-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Ulcer healing

SECONDARY OUTCOMES:
HIV viral load from genital ulcers
HIV viral load in semen

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Paz Bailey, MD, Principal Investigator — Centers for Disease Control and Prevention; David Lewis, MD, Principal Investigator — STIRC, National Institute for Communicable Diseases (NICD), South Africa
Locations (2):
- South Africa (2):
  - Eloff Street Clinic, Johannesburg, Gauteng
  - Green Door, Alexandra Health Centre, Johannesburg, Gauteng

REFERENCES:
- [Derived] Paz Bailey G, Sternberg M, Lewis DA, Puren A. Acute HIV infections among men with genital ulcer disease in South Africa. J Infect Dis. 2010 Jun 15;201(12):1811-5. doi: 10.1086/652785. PMID 20443734
- [Derived] Paz-Bailey G, Sternberg M, Puren AJ, Markowitz LE, Ballard R, Delany S, Hawkes S, Nwanyanwu O, Ryan C, Lewis DA. Improvement in healing and reduction in HIV shedding with episodic acyclovir therapy as part of syndromic management among men: a randomized, controlled trial. J Infect Dis. 2009 Oct 1;200(7):1039-49. doi: 10.1086/605647. PMID 19715417